CLINICAL TRIAL: NCT02938923
Title: Combining Testosterone Therapy and Exercise to Improve Function Post Hip Fracture
Brief Title: Starting a Testosterone and Exercise Program After Hip Injury
Acronym: STEP-HI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Maryland, Baltimore (Other); University of Colorado, Denver (Other); The University of Texas Medical Branch, Galveston (Other); Johns Hopkins University (Other); Harvard University (Other); University of Connecticut (Other); University of Utah (Other); University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Ellen F. Binder, MD, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AG051647 (NIH); 201609077 (Other: Washington University HRPO)
Record Dates: First submitted 2016-10-14; First posted 2016-10-19 (Estimated); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Hip Fracture; Frailty; Sarcopenia
MeSH Terms: conditions — Hip Fractures; Frailty; Sarcopenia | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and study staff conducting the interventions will be aware of the exercise group assignment. A Blinded Outcomes Assessor will be masked to study group assignment. Only the study pharmacist, an unblinded study physician, and Data Coordinating Center staff will be unblinded to gel treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Exercise + Testosterone (EX + T) (Experimental): Supervised exercise training 2 times per week and topical testosterone 1% gel (12.5 mg per pump depression) daily, both for six months duration.
  Interventions: Drug: Testosterone; Behavioral: Supervised exercise training
- Exercise + Placebo (EX + P) (Placebo Comparator): Supervised exercise training 2 times per week and placebo gel daily, both for six months duration.
  Interventions: Drug: Placebo gel; Behavioral: Supervised exercise training
- Enhanced Usual Care (EUC) (Other): Home exercise program 3 times per week and monthly health education modules, both for six months duration.
  Interventions: Behavioral: Home exercise program; Behavioral: Health Education Modules

INTERVENTIONS:
Drug: Testosterone — Topical testosterone gel 1%
  Other Names: T
  Arms: Exercise + Testosterone (EX + T)
Drug: Placebo gel — Inactive skin gel
  Other Names: P
  Arms: Exercise + Placebo (EX + P)
Behavioral: Supervised exercise training — Multicomponent exercise program focused primarily on progressive resistance exercise training
  Other Names: EX
  Arms: Exercise + Placebo (EX + P); Exercise + Testosterone (EX + T)
Behavioral: Home exercise program — Flexibility exercises performed at home 3 times per week and reviewed by study staff once a month.
  Other Names: EUC
  Arms: Enhanced Usual Care (EUC)
Behavioral: Health Education Modules — 30-40 minute presentations conducted by study staff for participants focused on health concerns unrelated to exercise.
  Other Names: EUC
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
This study is a randomized controlled double-blinded multi-center clinical trial enrolling female hip fracture patients who are 65 and older. It will compare the effects of six months of supervised exercise training combined with daily topical testosterone gel, to six months of supervised exercise and inactive gel, and to Enhanced Usual Care. The randomization protocol is that for every nine participants randomized, 4 will be assigned to the topical testosterone gel and supervised exercise training group; 4 will be assigned to topical inactive gel and supervised exercise training group; and 1 will be assigned to the enhanced usual care group. All participants will receive nutritional counseling, and calcium and vitamin D supplements.

DETAILED DESCRIPTION:
Hip fractures are common among older women and can have a devastating impact on their ability to remain independent. A clinically important functional decline and failure to recover following a hip fracture has been documented as late as a year after the fracture, even among women who were functioning at high levels before the event. Age-associated androgen deficiency in women contributes to deficits in muscle mass, strength and power that are common in this patient population before the fracture, and are exacerbated afterward. A pilot study of testosterone (T) supplementation in elderly female hip fracture patients has demonstrated the feasibility of T treatment in this population, and showed gains in lean body mass (LBM) and muscle strength with active drug, compared to placebo. The benefits of exercise in restoring muscle strength and physical function after a hip fracture have been documented. However, it remains unclear whether T treatment can augment the effects of exercise on mobility and patient-reported function after hip fracture.

The STEP-HI study is a 3-group, multi-center, randomized, placebo-controlled, double-blinded, parallel group clinical trial in older female hip fracture patients. Between 120 and 168 female hip fracture patients, age 65 years and older, will be randomized from multiple clinical sites in the USA, using objective screening criteria for T deficiency (serum total testosterone level < 60 ng/dL) and physical frailty (Modified Physical Performance Test (PPT) Score of 12-28). The primary study aim is to compare supervised exercise training (EX) with inactive (placebo) gel (EX+P) and EX combined with T therapy (EX+T), to ascertain the incremental impact of adding T to EX in older adult women with a recent hip fracture. The study team will carefully monitor testosterone levels, adverse events, biochemical parameters, and factors related to adherence to the interventions.

Information from this study has the potential to alter treatment of hip fracture in older women, a problem that contributes to significant morbidity and mortality, and has a large public health impact. The STEP-HI study is highly aligned with NIA's mission of identifying interventions that target common geriatric conditions and improve treatment options for older adults with multiple morbidities or risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Female 65 years and older.
* Surgical repair of a non-pathologic fracture of the proximal femur (Including: femoral neck or intracapsular, intertrochanteric, and subtrochanteric fractures) with a surgical repair date that is within 24 weeks at randomization. If a revision of such a fracture is performed due to failure of the repair, that surgery revision date may be used to calculate the time frame for the screening and randomization dates.
* Community-dwelling or in assisted living prior to the hip fracture event.
* Functional impairment at the time of screening, defined as a modified Physical Performance Score (mPPT) of 12-28.
* Serum total testosterone level <60 ng/dL.

Exclusion Criteria:

* Cognitive impairment or dementia of severity sufficient to interfere with ability to fully participate in the study or provide one's own informed consent, or a score of 11 or greater on the Short Blessed Test of Orientation, Memory and Concentration.
* Residence too far from research center (specific distance to be determined by each site) or planned travel greater than 2 weeks within the next 9 months.
* Anticipated to be permanently living in a nursing home at the time of randomization.
* Use of progestin or androgen containing compound within the previous 6 months.
* Treatment with systemic corticosteroids (daily dose > 5 mg prednisone or equivalent) for at least 90 days within the previous 12 months.
* Visual or hearing impairments that interfere with following directions for research procedures.
* Active or unstable cardiopulmonary disease (recent myocardial infarction, unstable angina, class III or IV Congestive Heart Failure) within prior 6 months, which would limit full participation in the study.
* Respiratory disease requiring chronic continuous oxygen therapy, or oxygen therapy during walking or exercise, which would limit full participation in this study.
* History of idiopathic deep venous thrombosis or pulmonary embolus (i.e., not related to period or immobilization or surgery), any pulmonary embolus less than 12 weeks prior to the first screening visit, recurrent or multiple venous thrombi; history of a hypercoagulable state such as Factor V Leiden thrombophilia.
* Musculoskeletal or neurological conditions that limit participation in this study, could be made worse by exercise training, or not expected to improve with exercise.
* Lower extremity amputation other than toes.
* Severe lower extremity pain or ulceration that could limit full participation in this study.
* History of: a) Breast, ovarian, endometrial or cervical cancer with diagnosis within the previous 10 years; b) Breast, ovarian, endometrial, or cervical cancer of Stage 2 or higher.
* History of HIV or active viral hepatitis.
* End Stage Renal Disease on dialysis or Glomerular Filtration Rate (GFR)<15 ml/min.
* Allergy to gel components.
* Recent history of alcohol or substance abuse, or current alcohol intake of ≥ 10 drinks/week.
* Planned joint surgery during the intervention period.
* Participation in another research study that in the site investigator's judgement could interfere or conflict with STEP-HI research assessments or interventions.
* Current use of aldactone, flutamide or leflunomide.
* Geriatric Depression Scale (GDS) score ≥ 12 at the screening assessment.
* Uncontrolled hypertension, defined as a systolic BP > 160 mmHg or diastolic BP > 95 mmHg, on at least two occasions.
* Elevated liver transaminase or alkaline phosphatase levels ≥ 2.5 times above normal range.
* Erythrocytosis defined as hematocrit > 51% (all sites but University of Utah) or ≥ 52% at University of Colorado - Denver and University of Utah sites.
* Severe anemia defined as Hgb < 7gm/dL.
* Uncontrolled diabetes defined as HgbA1C > 10%.
* Untreated or unstable thyroid disease, with serum Thyroid-stimulating Hormone (TSH) level ≥ 10 milli-international units per liter (mIU/L) or TSH level ≤ 0.4 mIU/L. Levels outside of the given range require site physician documentation addressing treatment or absence of thyroid disease and approval by the Central Coordinating Center (CCC).
* Site investigator's judgement that the participant would not be able to complete research procedures or interventions.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen F Binder, MD, Principal Investigator — Washington University School of Medicine; Kenneth B Schechtman, PhD, Principal Investigator — Washington University School of Medicine; Jay Magaziner, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (8):
- United States (8):
  - University of Colorado, Denver, Aurora, Colorado
  - University of Connecticut Heath - UConn Health, Farmington, Connecticut
  - University of Maryland School of Medicine/Johns Hopkins University, Baltimore, Maryland
  - HebrewSenior Life Harvard Medical School, Roslindale, Massachusetts
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch at Galveston (UTMB), Galveston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Binder EF, Christensen JC, Stevens-Lapsley J, Bartley J, Berry SD, Dobs AS, Fortinsky RH, Hildreth KL, Kiel DP, Kuchel GA, Marcus RL, McDonough CM, Orwig D, Sinacore DR, Schwartz RS, Volpi E, Magaziner J, Schechtman KB. A multi-center trial of exercise and testosterone therapy in women after hip fracture: Design, methods and impact of the COVID-19 pandemic. Contemp Clin Trials. 2021 May;104:106356. doi: 10.1016/j.cct.2021.106356. Epub 2021 Mar 11. PMID 33716173
- [Derived] Earp JE, Zhao S, Xu F, Kuo CL, Bartley JM, Fortinsky RH, Kositsawat J, Rehbein CO, Binder EF, Stevens-Lapsley J, Kuchel GA. Testosterone therapy effects adipose distribution in older females post hip-fracture: The STEP-HI study. Obes Pillars. 2026 Jan 12;17:100247. doi: 10.1016/j.obpill.2026.100247. eCollection 2026 Mar. PMID 41624165
- [Derived] Binder EF, Bartley JM, Berry SD, Dore PM, Fisher SR, Fortinsky RH, Guild C, Kiel DP, Kuchel GA, Marcus RL, McDonough CM, Monroe KM, Orwig DL, Paluch RA, Reeds D, Stevens-Lapsley J, Volpi E, Schechtman KB, Magaziner JS. Combining Exercise Training and Testosterone Therapy in Older Women After Hip Fracture: The STEP-HI Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e2510512. doi: 10.1001/jamanetworkopen.2025.10512. PMID 40372752
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2018 and February 2023, participants identified from hospital records or referred from physicians/rehabilitation staff at 8 academic medical centers, were approached 6-24 weeks following hip repair surgery. If eligible by chart review, participants were pre-screened, consented for full study, screened, and completed baseline assessments, prior to randomization. The first participant was randomized in March 2019 and the final participant randomized in February 2023.
Pre-assignment Details: 4695 charts were reviewed. 907 were eligible by chart review and 344 agreed to complete the pre-screening questionnaire. Of those, 28 failed, another 42 were deemed ineligible after further review, 7 refused to review the consent, and 60 refused consent. Leaving 207 who consented for screening, of which 12 refused to continue to screening visit and 10 were found ineligible prior to screening. 185 screened, of whom 32 screen failed, 7 refused after screening, and 17 were ineligible to randomize.
Groups:
- Exercise + Testosterone (EX + T): Supervised exercise training 2 times per week and topical testosterone 1% gel (12.5 mg per pump depression), both for six months duration.
  Testosterone: Topical testosterone gel 1%
  Supervised exercise training: Multicomponent exercise program focused primarily on progressive resistance exercise training
Period: Overall Study
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC)
Started | 55 | 54 | 20
Completed | 54 | 51 | 19
Not Completed | 1 | 3 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC) | Total
Number analyzed (Participants) | 55 | 54 | 20 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.42 (9.08) | 78.28 (7.52) | 82.98 (8.39) | 79.49 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 54 | 20 | 129
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 1 | 5
  Not Hispanic or Latino | 54 | 48 | 18 | 120
  Unknown or Not Reported | 0 | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 1 | 6
  White | 52 | 49 | 19 | 120
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 55 | 54 | 20 | 129
Site [Count of Participants; unit: Participants]
  Hebrew SeniorLife (HSL)/Beth Israel (BI)/Harvard Medical School | 17 | 16 | 5 | 38
  Washington University in St. Louis (WashU) | 9 | 12 | 5 | 26
  University of Colorado - Denver (UCD) | 1 | 0 | 2 | 3
  University of Connecticut (UConn Health) | 11 | 11 | 4 | 26
  University of Maryland Baltimore/Johns Hopkins University (UM/JH) | 1 | 0 | 2 | 3
  University of Texas Medical Branch at Galveston (UTMB) | 8 | 7 | 1 | 16
  University of Utah Health (UofU) | 5 | 4 | 0 | 9
  University of Pittsburgh (Pitt)/University of Pittsburgh Medical Center (UPMC) | 3 | 4 | 1 | 8
Time from hip surgery to baseline start date [Mean (Standard Deviation); unit: days] | 98.29 (32.52) | 108.54 (33.42) | 89.65 (21.62) | 101.24 (32.02)
Type of Fracture [Count of Participants; unit: Participants]
  Intertrochanteric Fracture | 23 | 23 | 13 | 59
  Intracapsular or Femoral Neck Fracture | 25 | 22 | 3 | 50
  Subtrochanteric Fracture | 7 | 9 | 4 | 20
Body mass index (BMI) [Median (Standard Deviation); unit: Kilograms/meters ^2 (kg/m^2)] | 25.61 (5.49) | 26.89 (5.02) | 24.43 (3.36) | 25.96 (5.06)
History of Lung Disease [Count of Participants; unit: Participants]
  No lung disease | 51 | 51 | 16 | 118
  lung disease | 4 | 3 | 4 | 11
Co-morbidity count [Mean (Standard Deviation); unit: units on a scale] — Individual co-morbidities from the STEP-HI Medical Health Questionnaire were counted giving each participant a score ranging from 0 to 38. A score of 0 represents no co-morbidities and a score of 38 represents having all counted diagnoses.
  units on a scale | 5.20 (3.09) | 5.13 (2.52) | 5.85 (3.17) | 5.27 (2.86)
Geriatric Depression Scale (GDS) [Mean (Standard Deviation); unit: unites on a scale] — The Geriatric Depression Scale short form is a standardized, self-report measure of depression validated for older adults. The scale contains 15 yes or no items. Scores range from 0 to 15. Scores of 0 to 5 are considered normal, while scores greater than 5 suggest depression. The higher the score, the more severe the depression.
  unites on a scale | 1.84 (1.75) | 2.43 (2.04) | 3.15 (2.62) | 2.29 (2.06)
Six Minute Walk Distance [Mean (Standard Deviation); unit: meters] — Walking endurance was measured using a 6-Minute Walk Distance. Participants were asked to walk back and forth on a measured path marked clearly at both ends for turning purposes, while being told when each minute has passed, and receiving verbal encouragement every 60 seconds. Total distance was measured in meters with higher distances equating to higher walking endurance.
  meters | 267.77 (86.60) | 225.92 (98.09) | 206.37 (76.82) | 240.73 (92.82)
Total lean body mass [Mean (Standard Deviation); unit: Grams] — Total lean body mass measured by dual x-ray absorptiometry (DXA). Baseline DXA scans were completed prior to the first administration of study drug. All scans were completed prior to exercise or 1-RM measurements if scheduled for the same day. DXA scans were reviewed for quality control, proper positioning, and artifacts centrally.
  Grams | 36649.42 (5892.42) | 37744.01 (5543.42) | 35144.55 (4276.92) | 36874.31 (5558.35)
Appendicular lean body mass [Mean (Standard Deviation); unit: Grams] — Lean body mass of the arms and legs, measured by dual x-ray absorptiometry (DXA). Baseline DXA scans were completed prior to the first administration of study drug. All scans were completed prior to exercise or 1-RM measurements if scheduled for the same day. DXA scans were reviewed for quality control, proper positioning, and artifacts centrally.
  Grams | 15650.59 (3045.80) | 16276.07 (3078.32) | 15070.01 (2279.41) | 15822.42 (2965.91)
Leg Press 1-Repetition Maximum [Mean (Standard Deviation); unit: Pounds] — Muscle strength measured as the maximal amount of weight that the participant was able to lift for one repetition (1-RM). The 1-RM is defined as the greatest resistance that could be overcome through a defined range of motion using proper techniques. 1-RM was obtained using the fractured and unfractured legs simultaneously, on identical inclined leg press machines (Inflight model CT-ILPC) across clinical sites. Subjects were asked to move against progressively heavier resistance loads until a repetition failure was achieved. A rest period separated each increase in weight. Population: 7 participants attempted, but were unable to complete the 1-RM (unable to move the weight at all) and 2 participants refused to attempt the measure.
  Pounds
    number analyzed (Participants) | 53 | 49 | 18 | 120
    (all) | 97.12 (53.86) | 85.41 (40.97) | 88.61 (55.16) | 91.06 (49.09)
Modified Physical Performance (mPPT) Score [Mean (Standard Deviation); unit: units on a scale] — A modified version of the Physical Performance Test (mPPT) was used to measure physical function. Participants were asked to complete 9 standardized tasks (book lift, putting on a lab coat, picking up a penny from the floor, standing balance, standing up five times from a 16-inch chair, 50 foot walk including a turn, 360 degree turn, stair climb for 10 steps, and climbing 2 additional flights of steps) for a total score ranging from 0 (significant impairment) to 36 (excellent functioning).
  units on a scale | 20.85 (6.73) | 20.37 (6.84) | 17.55 (6.95) | 20.14 (6.85)
Short Physical Performance Battery (SPPB) [Mean (Standard Deviation); unit: units on a scale] — The Short Physical Performance Battery (SPPB) is a well validated objective physical performance measure used to identify risk for disability. The SPPB consists of 3 tasks: chair rise, progressive Romberg balance, and gait speed on a 4 meter walk (both at preferred normal speed and fast pace). Each task was scored (0-4) with a total range of 0 to 12. Participants who score 0 are unable to complete the tasks and participants with higher scores are considered to have higher functional mobility.
  units on a scale | 6.95 (2.16) | 6.63 (2.27) | 5.45 (2.14) | 6.58 (2.25)
Older Adult Resources and Services (OARS) Activities of Daily Living (ADL) Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Duke Older Adult Resources and Services (OARS) Multidimensional Functional Assessment Questionnaire complete Activities of Daily Living (ADL) is a standardized, valid and reliable, self-report questionnaire used to determine the effect of services on the functional status of older adults. The respondents were asked about their ability to perform basic (BADL) and instrumental (IADL) activities of daily living. The OARS basic and instrumental ALD subscales are both measured by 7 questions with scores from 0 (meaning significant impairment) to 14 (meaning excellent functioning).
  units on a scale
    Basic Activities of Daily Living (BADL) | 12.15 (1.67) | 12.0 (2.01) | 12.05 (1.76) | 12.07 (1.82)
    Instrumental Activities of Daily Living (IADL) | 11.51 (2.43) | 11.28 (2.48) | 11.35 (1.93) | 11.39 (2.37)
Functional Status Questionnaire (FSQ) [Mean (Standard Deviation); unit: units on a scale] — The Functional Status Questionnaire (FSQ) is a self-reported measure asking about the amount of difficulty a participant experienced when performing daily tasks in the previous 4 weeks. There are a total of 6 subscales, but only the basic ADL and Intermediate ADL were used in the STEP-HI study for a total of 9 items. Scores range from 0 (high amount of difficulty completing tasks) to 36 (no difficulty completing tasks).
  units on a scale | 23.16 (4.80) | 21.80 (5.03) | 21.30 (5.15) | 22.30 (4.97)
Hip Rating Questionnaire (HRQ) [Mean (Standard Deviation); unit: units on a scale] — The Hip Rating Questionnaire (HRQ) Standardized is a 14-item scale with weighted questions regarding quality of life (pain level and ability to walk) and function (ability to use stairs, put on socks/shoes, use public transportation, bathe, shop, do housework, and get in and out of a chair/bed) related to the hip fracture event. The scale scores range from 16 to 100. Higher scores are associated with less pain, higher function, and better quality of life.
  units on a scale | 72.06 (12.36) | 69.54 (10.227) | 70.89 (11.87) | 70.82 (11.42)
Bone mineral density (BMD) of non-fractured proximal femur [Mean (Standard Deviation); unit: Grams/centimeters^2 (g/cm^2)] — Bone mineral density (BMD) measured by dual x-ray absorptiometry (DXA) of the non-fractured proximal femur in participants without hardware in the contralateral hip. Baseline DXA scans were completed prior to the first administration of study drug. All scans were completed prior to exercise or 1-RM measurements if scheduled for the same day. DXA scans were reviewed for quality control, proper positioning, and artifacts centrally. Population: Only participants without hardware in their contralateral hip (opposite hip to the surgical repair conducted just prior to enrollment in the STEP-HI study) completed the DXA scan for BMD. A total of 9 EX+T, 6 EX+P, and 4 EUC participants were not scanned.
  Grams/centimeters^2 (g/cm^2)
    number analyzed (Participants) | 46 | 48 | 16 | 110
    (all) | 0.71 (0.12) | 0.73 (0.12) | 0.71 (0.12) | 0.72 (0.12)
Patient-Reported Outcomes Measurement Information System (PROMIS®) Global Health [Mean (Standard Deviation); unit: T-score] — Patient-Reported Outcomes Measurement Information System (PROMIS®) Global Health instrument is a 10 item self report questionnaire used to measure overall quality of life using 2 summary scores: physical and mental health. PROMIS® Global Health was developed and validated to be psychometrically accurate for the general population, as well as individuals with chronic conditions. Each summary score is standardized to the general population, with the average T-score for the US population being 50 and standard deviation of 10. Higher scores represent better global health.
  T-score
    Mental Health T-score | 51.75 (6.20) | 51.07 (6.39) | 47.75 (7.99) | 50.84 (6.67)
    Physical Health T-score | 48.29 (6.35) | 46.21 (6.51) | 45.59 (5.99) | 47.00 (6.42)
Serum Testosterone Level (Total) [Mean (Standard Deviation); unit: nanograms per deciliter (ng/dL)] — Serum total testosterone as measured by liquid chromatography - tandem mass spectrometry (LC-MS) test methodology. Total testosterone levels under 7.0 ng/dL are not detectable. In these cases, 6.9 was used in place of a missing value.
  nanograms per deciliter (ng/dL) | 15.67 (9.19) | 17.24 (12.50) | 13.02 (5.85) | 15.92 (10.37)
Serum Testosterone Level (Free) [Mean (Standard Deviation); unit: nanograms per deciliter (ng/dL)] — Serum free testosterone as measured by liquid chromatography - tandem mass spectrometry (LC-MS) test methodology. The lowest value of free testosterone which was detectable was 1.12. Lab reports with undetectably low values were set to 1.12. Population: The central lab was unable to process free testosterone for certain periods due to equipment failure. The measurement was obtained if possible.
  nanograms per deciliter (ng/dL)
    number analyzed (Participants) | 37 | 32 | 17 | 86
    (all) | 0.24 (0.18) | 0.25 (0.14) | 0.17 (0.09) | 0.22 (0.15)
Hand grip strength - left hand [Mean (Standard Deviation); unit: Kilograms (kg)] — Hand grip strength measured by hand dynamometer to obtain the average of 3 trials. Population: One participant was unable to preform the hand grip in the left hand.
  Kilograms (kg)
    number analyzed (Participants) | 54 | 54 | 20 | 128
    (all) | 15.27 (6.04) | 15.96 (5.49) | 15.82 (5.45) | 15.65 (5.68)
Hand grip strength - right hand [Mean (Standard Deviation); unit: Kilograms (kg)] — Hand grip strength measured by hand dynamometer to obtain the average of 3 trials.
  Kilograms (kg) | 16.45 (5.84) | 17.44 (5.95) | 16.95 (5.69) | 16.95 (5.84)

OUTCOME MEASURES:

1. Primary Outcome: Change in Six Minute Walk Distance
Description: Walking endurance was measured using a 6-Minute Walk Distance. Participants were asked to walk back and forth on a measured path marked clearly at both ends for turning purposes, while being told when each minute has passed, and receiving verbal encouragement every 60 seconds. Total distance was measured in meters with higher distances equating to higher walking endurance. Each individual participant distance from Baseline was subtracted from Month 6 to represent change over the length of the study. Higher positive values represent more improvement in walking distance. In addition to the primary analysis (unadjusted baseline to 6 month comparison), statistical contracts were evaluated to determine if there was significant between-group differences in the change from baseline to 3 months and additional analysis of covariance were performed to adjust for baseline values and covariates that differed across groups at baseline.
Time Frame: Baseline to 6 months
Population: Randomized participants (N=122) who completed the primary outcome measure at baseline and one other follow-up time point (3 Months or 6 Months post randomization).
Measure: Least Squares Mean (95% Confidence Interval); unit: Meters
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 53 | 51 | 18
Meters
  Unadjusted baseline to 6 months | 42.69 [26.35 to 59.04] | 40.50 [23.82 to 57.18] | 37.65 [8.29 to 67.02]
  Baseline to 6 month with covariates | 42.38 [24.96 to 59.80] | 41.75 [23.98 to 59.52] | 33.95 [4.30 to 63.60]
  Unadjusted baseline to 3 months | 24.10 [9.72 to 38.48] | 29.18 [14.37 to 43.99] | 37.60 [12.00 to 63.20]
  Baseline to 3 months with covariates | 24.72 [11.87 to 37.56] | 30.23 [16.98 to 43.48] | 38.36 [15.76 to 60.96]
Statistical Analysis 1: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to six months from mixed model ANOVA with an unstructured covariance structure; Test type: Superiority; p = 0.853, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 0.19; Mean Difference (Final Values) = 2.19, 95% CI 2-sided [-21.16 to 25.54] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 2: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.767, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 0.30; Mean Difference (Final Values) = 5.04, 95% CI 2-sided [-28.57 to 38.65] — Difference between the changes (EX+T - EUC)
Statistical Analysis 3: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.868, Mixed Models Analysis — Unadjusted p-value; t (df,112) = 0.17; Mean Difference (Final Values) = 2.84, 95% CI 2-sided [-30.93 to 36.62] — Difference between the changes (EX+P - EUC)
Statistical Analysis 4: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to six months from mixed model ANOVA with a Toeplitz covariance structure in the model with covariates; Test type: Superiority; p = 0.960, Mixed Models Analysis — Unadjusted p-value; t (df, 217) = 0.05; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-24.26 to 25.52] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 5: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.630, Mixed Models Analysis — Unadjusted p-value; t (df, 217) = 0.48; Mean Difference (Final Values) = 8.42, 95% CI 2-sided [-25.97 to 42.82] — Difference between the changes (EX+T - EUC)
Statistical Analysis 6: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.657, Mixed Models Analysis — Unadjusted p-value; t (df, 217) = 0.44; Mean Difference (Final Values) = 7.79, 95% CI 2-sided [-26.77 to 42.36] — Difference between the changes (EX+P - EUC)
Statistical Analysis 7: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to three months from mixed model ANOVA with an unstructured covariance structure; Test type: Superiority; p = 0.627, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -0.49; Mean Difference (Final Values) = -5.08, 95% CI 2-sided [-25.72 to 15.56] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 8: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.364, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -0.91; Mean Difference (Final Values) = -13.50, 95% CI 2-sided [-42.86 to 15.86] — Difference between the changes (EX+T - EUC)
Statistical Analysis 9: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.574, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -0.56; Mean Difference (Final Values) = -8.42, 95% CI 2-sided [-38.00 to 21.15] — Difference between the changes (EX+P - EUC)
Statistical Analysis 10: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to three months from mixed model ANOVA with a Toeplitz covariance structure in the model with covariates; Test type: Superiority; p = 0.557, Mixed Models Analysis — Unadjusted p-value; t (df, 217) = -0.59; Mean Difference (Final Values) = -5.51, 95% CI 2-sided [-23.96 to 12.94] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 11: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 10]; Test type: Superiority; p = 0.302, Mixed Models Analysis — Unadjusted p-value; t (df, 217) = -1.03; Mean Difference (Final Values) = -13.65, 95% CI 2-sided [-39.64 to 12.35] — Difference between the changes (EX+T - EUC)
Statistical Analysis 12: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 10]; Test type: Superiority; p = 0.541, Mixed Models Analysis — Unadjusted p-value; t (df, 217) = -0.61; Mean Difference (Final Values) = -8.14, 95% CI 2-sided [-34.33 to 18.06] — Difference between the changes (EX+P - EUC)

2. Secondary Outcome: Change in Total Lean Body Mass
Description: Total lean body mass measured by dual x-ray absorptiometry (DXA). Baseline DXA scans were completed prior to the first administration of study drug. All scans were completed prior to exercise or 1-RM measurements if scheduled for the same day. DXA scans were reviewed for quality control, proper positioning, and artifacts centrally. Each individual participant measure from Baseline was subtracted from Month 6 to represent change over the length of the study. Higher positive values represent more gains in total lean body mass. Per the protocol: In addition to the primary analysis (unadjusted baseline to 6 month comparison), additional analysis of covariance were performed to adjust for baseline values and covariates that differed across groups at baseline. DXA was not performed at 3 months.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: grams
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 53 | 51 | 18
grams
  Unadjusted baseline to 6 month | 922.91 [414.98 to 1430.83] | 565.19 [36.04 to 1094.33] | -14.02 [-972.19 to 944.14]
  Baseline to 6 month with covariates | 930.80 [480.76 to 1380.83] | 547.43 [79.29 to 1015.57] | 94.16 [-689.19 to 877.50]
Statistical Analysis 1: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.336, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 0.97; Mean Difference (Final Values) = 357.72, 95% CI 2-sided [-375.75 to 1091.19] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 2: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.090, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 1.71; Mean Difference (Final Values) = 936.93, 95% CI 2-sided [-147.56 to 2021.42] — Difference between the changes (EX+T - EUC)
Statistical Analysis 3: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.297, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 1.05; Mean Difference (Final Values) = 579.21, 95% CI 2-sided [-515.36 to 1673.78] — Difference between the changes (EX+P - EUC)
Statistical Analysis 4: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to six months from mixed model ANOVA with a Heterogeneous Toeplitz covariance structure in the model with covariates; Test type: Superiority; p = 0.245, Mixed Models Analysis — Unadjusted p-value; t (df, 107) = 1.17; Mean Difference (Final Values) = 383.36, 95% CI 2-sided [-266.06 to 1032.79] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 5: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.069, Mixed Models Analysis — Unadjusted p-value; t (df, 107) = 1.84; Mean Difference (Final Values) = 836.64, 95% CI 2-sided [-67.04 to 1740.32] — Difference between the changes (EX+T - EUC)
Statistical Analysis 6: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.327, Mixed Models Analysis — Unadjusted p-value; t (df, 107) = 0.98; Mean Difference (Final Values) = 453.28, 95% CI 2-sided [-459.13 to 1365.68] — Difference between changes (EX+P - EUC)

3. Secondary Outcome: Change in Appendicular Lean Body Mass
Description: Lean body mass of the arms and legs, measured by dual x-ray absorptiometry (DXA). Baseline DXA scans were completed prior to the first administration of study drug. All scans were completed prior to exercise or 1-RM measurements if scheduled for the same day. DXA scans were reviewed for quality control, proper positioning, and artifacts centrally. Each individual participant measure from Baseline was subtracted from Month 6 to represent change over the length of the study. Higher positive values represent more gains in appendicular lean body mass. Per the protocol: In addition to the primary analysis (unadjusted baseline to 6 month comparison), additional analysis of covariance were performed to adjust for baseline values and covariates that differed across groups at baseline. DXA was not performed at 3 months.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: grams
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 53 | 51 | 18
grams
  Unadjusted baseline to 6 month | 446.35 [163.20 to 729.49] | 429.19 [134.19 to 724.20] | -116.29 [-650.56 to 417.97]
  Baseline to 6 month with covariates | 453.30 [176.93 to 729.66] | 419.57 [131.61 to 707.53] | -212.45 [-699.35 to 274.44]
Statistical Analysis 1: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.934, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 0.08; Mean Difference (Final Values) = 17.16, 95% CI 2-sided [-391.74 to 426.05] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 2: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.068, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 1.84; Mean Difference (Final Values) = 562.64, 95% CI 2-sided [-42.02 to 1167.31] — Difference between the changes (EX+T - EUC)
Statistical Analysis 3: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.079, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 1.77; Mean Difference (Final Values) = 545.49, 95% CI 2-sided [-64.81 to 1155.79] — Difference between the changes (EX+P - EUC)
Statistical Analysis 4: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to six months from mixed model ANOVA with an unstructured covariance structure in the model with covariates; Test type: Superiority; p = 0.867, Mixed Models Analysis — Unadjusted p-value; t (df, 102) = 0.17; Mean Difference (Final Values) = 33.73, 95% CI 2-sided [-365.40 to 432.860] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 5: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.020, Mixed Models Analysis — Unadjusted p-value; t (df, 102) = 2.36; Mean Difference (Final Values) = 665.75, 95% CI 2-sided [105.68 to 1225.81] — Difference between the changes (EX+T - EUC)
Statistical Analysis 6: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.029, Mixed Models Analysis — Unadjusted p-value; t (df, 102) = 2.22; Mean Difference (Final Values) = 632.02, 95% CI 2-sided [66.38 to 1197.66] — Difference between the changes (EX+P - EUC)

4. Secondary Outcome: Change in 1-repetition Maximum (1-RM) Leg Press Strength
Description: Muscle strength measured as the maximal amount of weight that the participant was able to lift for one repetition (1-RM). The 1-RM is defined as the greatest resistance that could be overcome through a defined range of motion using proper techniques. Subjects were asked to move against progressively heavier resistance loads until a repetition failure was achieved. Each individual participant measure from Baseline was subtracted from Month 6 to represent change over the length of the study. Higher positive values represent the increased ability to lift more weight. Per the protocol: In addition to the primary analysis (unadjusted baseline to 6 month comparison), statistical contracts were evaluated to determine if there was significant between-group differences in the change from baseline to 3 months and additional analysis of covariance were performed to adjust for baseline values and covariates that differed across groups at baseline.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: pounds
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 53 | 51 | 18
pounds
  Unadjusted baseline to 6 month | 62.62 [48.50 to 76.73] | 61.91 [47.32 to 76.51] | 38.18 [13.20 to 63.16]
  Baseline to 6 month with covarites | 64.26 [50.78 to 77.74] | 59.45 [45.37 to 73.54] | 39.36 [15.86 to 62.85]
  Unadjusted baseline to 3 month | 38.71 [28.81 to 48.60] | 40.09 [29.73 to 50.45] | 23.23 [5.50 to 40.96]
  Baseline to 3 month with covariates | 39.01 [29.77 to 48.25] | 39.25 [29.54 to 48.95] | 24.52 [7.87 to 41.17]
Statistical Analysis 1: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.946, Mixed Models Analysis — Unadjusted p-value; t (df, 110) = 0.07; Mean Difference (Final Values) = 0.70, 95% CI 2-sided [-19.61 to 21.01] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 2: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.094, Mixed Models Analysis — Unadjusted p-value; t (df, 110) = 1.69; Mean Difference (Final Values) = 24.44, 95% CI 2-sided [-4.25 to 53.13] — Difference between the changes (EX+T - EUC)
Statistical Analysis 3: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.107, Mixed Models Analysis — Unadjusted p-value; t (df, 110) = 1.63; Mean Difference (Final Values) = 23.74, 95% CI 2-sided [-5.19 to 52.67] — Difference between the changes (EX+P - EUC)
Statistical Analysis 4: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.627, Mixed Models Analysis — Unadjusted p-value; t (df, 189) = 0.49; Mean Difference (Final Values) = 4.81, 95% CI 2-sided [-14.68 to 24.30] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 5: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.072, Mixed Models Analysis — Unadjusted p-value; t (df, 189) = 1.81; Mean Difference (Final Values) = 24.91, 95% CI 2-sided [-2.20 to 52.01] — Difference between the changes (EX+T - EUC)
Statistical Analysis 6: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.149, Mixed Models Analysis — Unadjusted p-value; t (df, 189) = 1.45; Mean Difference (Final Values) = 20.10, 95% CI 2-sided [-7.29 to 47.49] — Difference between the changes (EX+P - EUC)
Statistical Analysis 7: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.849, Mixed Models Analysis — Unadjusted p-value; t (df, 110) = -0.19; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-15.71 to 12.95] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 8: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.134, Mixed Models Analysis — Unadjusted p-value; (df, 110) = 1.15; Mean Difference (Final Values) = 15.47, 95% CI 2-sided [-4.83 to 35.78] — Difference between the changes (EX+T - EUC)
Statistical Analysis 9: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.107, Mixed Models Analysis — Unadjusted p-value; t (df, 110) = 1.63; Mean Difference (Final Values) = 16.86, 95% CI 2-sided [-3.68 to 37.39] — Difference between the changes (EX+P - EUC)
Statistical Analysis 10: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 1, analysis 10]; Test type: Superiority; p = 0.973, Mixed Models Analysis — Unadjusted p-value; t (df, 189) = -0.03; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-13.64 to 13.17] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 11: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 10]; Test type: Superiority; p = 0.135, Mixed Models Analysis — Unadjusted p-value; t (df, 189) = 1.50; Mean Difference (Final Values) = 14.49, 95% CI 2-sided [-4.56 to 33.54] — Difference between the changes (EX+T - EUC)
Statistical Analysis 12: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 10]; Test type: Superiority; p = 0.134, Mixed Models Analysis — Unadjusted p-value; t (df, 189) = 1.51; Mean Difference (Final Values) = 14.72, 95% CI 2-sided [-4.55 to 34.00] — Difference between the changes (EX+P - EUC)

5. Secondary Outcome: Change in Total Modified Physical Performance Test (mPPT) Score
Description: A modified version of the Physical Performance Test (mPPT) was used to measure physical function. Participants were asked to complete 9 standardized tasks (book lift, putting on a lab coat, picking up a penny from the floor, standing balance, standing up five times from a 16-inch chair, 50 foot walk including a turn, 360 degree turn, stair climb for 10 steps, and climbing 2 additional flights of steps) for a total score ranging from 0 (significant impairment) to 36 (excellent functioning). Each individual participant score from Baseline was subtracted from Month 6 to represent change over the length of the study. Higher positive values represent more improvement in physical functioning.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 53 | 51 | 18
units on a scale
  Unadjusted baseline to 6 month | 3.32 [2.24 to 4.41] | 2.12 [1.01 to 3.22] | 2.97 [1.00 to 4.95]
  baseline to 6 month with covariates | 3.33 [2.03 to 4.64] | 2.20 [0.87 to 3.52] | 2.74 [0.53 to 4.95]
  Unadjusted baseline to 3 month | 2.60 [1.55 to 3.64] | 1.12 [0.04 to 2.19] | 2.26 [0.40 to 4.11]
  Baseline to 3 month with covariates | 2.61 [1.69 to 3.54] | 1.15 [0.20 to 2.11] | 2.31 [0.70 to 3.93]
Statistical Analysis 1: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.125, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 1.55; Mean Difference (Final Values) = 1.21, 95% CI 2-sided [-0.34 to 2.76] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 2: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.758, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 0.31; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-1.90 to 2.61] — Difference between the changes (EX+T - EUC)
Statistical Analysis 3: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.455, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -0.75; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-3.12 to 1.41] — Difference between the changes (EX+P - EUC)
Statistical Analysis 4: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.229, Mixed Models Analysis — Unadjusted p-value; t (df, 214) = 1.21; Mean Difference (Final Values) = 1.14, 95% CI 2-sided [-0.72 to 3.00] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 5: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.647, Mixed Models Analysis — Unadjusted p-value; t (df, 214) = 0.46; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [-1.97 to 3.16] — Difference between the changes (EX+T - EUC)
Statistical Analysis 6: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.680, Mixed Models Analysis — Unadjusted p-value; t (df, 214) = -0.41; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-3.12 to 2.04] — Difference between the changes (EX+P - EUC)
Statistical Analysis 7: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.052, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 1.96; Mean Difference (Final Values) = 1.48, 95% CI 2-sided [-0.02 to 2.97] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 8: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.754, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 0.31; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-1.79 to 2.46] — Difference between the changes (EX+T - EUC)
Statistical Analysis 9: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.294, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -1.06; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-3.28 to 1.00] — Difference between the changes (EX+P - EUC)
Statistical Analysis 10: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to three months from mixed model ANOVA with an unstructured covariance structure in the model with covariates; Test type: Superiority; p = 0.031, Mixed Models Analysis — Unadjusted p-value; t (df, 214) = 2.17; Mean Difference (Final Values) = 1.46, 95% CI 2-sided [0.13 to 2.78] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 11: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 5, analysis 10]; Test type: Superiority; p = 0.752, Mixed Models Analysis — Unadjusted p-value; t (df, 214) = 0.32; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-1.56 to 2.16] — Difference between the changes (EX+T - EUC)
Statistical Analysis 12: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 5, analysis 10]; Test type: Superiority; p = 0.223, Mixed Models Analysis — Unadjusted p-value; t (df, 214) = -1.22; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-3.03 to 0.71] — Difference between the changes (EX+P - EUC)

6. Secondary Outcome: Change in Short Physical Performance Battery (SPPB) Score
Description: The Short Physical Performance Battery (SPPB) is a well validated objective physical performance measure used to identify risk for disability. The SPPB consists of: chair rise, progressive Romberg balance, and 4 meter gait speed. Each task was scored (0-4) with a total range of 0-12. Participants who score 0 are unable to complete the tasks and participants with higher scores are considered to have higher functional mobility. Each individual participant score from Baseline was subtracted from Month 6 to represent change over the length of the study. Higher positive values represent more improvement in physical performance. In addition to the primary analysis (unadjusted baseline to 6 month comparison), statistical contracts were evaluated to determine if there was significant between-group differences in the change from baseline to 3 months and additional analysis of covariance were performed to adjust for baseline values and covariates that differed across groups at baseline.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 53 | 51 | 18
units on a scale
  Unadjusted baseline to 6 month | 1.53 [1.11 to 1.96] | 0.68 [0.25 to 1.11] | 1.45 [0.67 to 2.24]
  Baseline to 6 month with covariates | 1.55 [1.12 to 1.99] | 0.73 [0.29 to 1.17] | 1.43 [0.65 to 2.21]
  Unadjusted baseline to 3 month | 1.02 [0.59 to 1.45] | 0.32 [-0.12 to 0.77] | 1.11 [0.35 to 1.88]
  Baseline to 3 month with covariates | 1.03 [0.66 to 1.40] | 0.35 [-0.03 to 0.74] | 1.11 [0.44 to 1.77]
Statistical Analysis 1: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.006, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 2.78; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [0.24 to 1.46] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 2: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.863, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 0.17; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.81 to 0.97] — Difference between the changes (EX+T - EUC)
Statistical Analysis 3: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.091, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -1.71; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-1.67 to 0.12] — Difference between the changes (EX+P - EUC)
Statistical Analysis 4: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to six months from mixed model ANOVA with an Autoregressive (1) covariance structure in the model with covariates; Test type: Superiority; p = 0.009, Mixed Models Analysis — Unadjusted p-value; t (df, 214) = 2.65; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [0.21 to 1.44] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 5: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p = 0.778, Mixed Models Analysis — Unadjusted p-value; t (df, 214) = 0.28; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.76 to 1.02] — Difference between the changes (EX+T - EUC)
Statistical Analysis 6: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p = 0.124, Mixed Models Analysis — Unadjusted p-value; t (df, 214) = -1.55; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.59 to 0.19] — Difference between the changes (EX+P - EUC)
Statistical Analysis 7: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.027, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 2.24; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [0.08 to 1.31] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 8: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.833, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -0.21; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.97 to 0.78] — Difference between the changes (EX+T - EUC)
Statistical Analysis 9: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.080, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -1.77; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-1.67 to 0.10] — Difference between the changes (EX+P - EUC)
Statistical Analysis 10: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to three months from mixed model ANOVA with an Autoregressive (1) covariance structure in the model with covariates; Test type: Superiority; p = 0.014, Mixed Models Analysis — Unadjusted p-value; t (df, 214) = 2.49; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [0.14 to 1.21] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 11: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 6, analysis 10]; Test type: Superiority; p = 0.834, Mixed Models Analysis — Unadjusted p-value; t (df, 214) = -0.21; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.84 to 0.68] — Difference between the changes (EX+T - EUC)
Statistical Analysis 12: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 6, analysis 10]; Test type: Superiority; p = 0.054, Mixed Models Analysis — Unadjusted p-value; t (df, 214) = -1.94; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.52 to 0.01] — Difference between the changes (EX+P - EUC)

7. Secondary Outcome: Change in Older Adult Resources and Services (OARS) Activities of Daily Living (ADL) Questionnaire
Description: The OARS Multidimensional Functional Assessment Questionnaire Activities of Daily Living (ADL) is a standardized, valid and reliable, self-report questionnaire used to determine the effect of services on the functional status of older adults by asking respondents about their ability to perform ADLS on 2 subscales: Basic (BADL) and Instrumental (IADL). Both subscales are scored from 0 (significant impairment) to 14 (excellent functioning). The individual participant score from Baseline was subtracted from Month 6 to represent change over the length of the study. Higher positive values represent more improvement in functioning. In addition to the primary analysis (unadjusted baseline to 6 month comparison), statistical contracts were evaluated to determine if there was significant between-group differences in the change from baseline to 3 months and additional analysis of covariance were performed to adjust for baseline values and covariates that differed across groups at baseline.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 53 | 51 | 18
units on a scale
  BADL Unadjusted baseline to 6 month | 0.60 [0.25 to 0.94] | 0.35 [0.00 to 0.71] | 0.79 [0.20 to 1.37]
  BADL Baseline to 6 month with covariates | 0.59 [0.20 to 0.98] | 0.36 [-0.04 to 0.75] | 0.83 [0.19 to 1.48]
  BADL Unadjusted baseline to 3 month | 0.36 [0.03 to 0.69] | 0.14 [-0.20 to 0.47] | 0.56 [-0.03 to 1.15]
  BADL Baseline to 3 month with covariates | 0.36 [0.04 to 0.68] | 0.14 [-0.19 to 0.47] | 0.59 [0.02 to 1.16]
  IADL Unadjusted baseline to 6 month | 0.39 [-0.05 to 0.82] | 0.51 [0.07 to 0.94] | 0.81 [0.08 to 1.54]
  IADL Baseline to 6 month with covariates | 0.40 [-0.03 to 0.82] | 0.51 [0.08 to 0.95] | 0.74 [0.04 to 1.45]
  IADL Unadjusted baseline to 3 month | 0.70 [0.33 to 1.07] | 0.47 [0.09 to 0.85] | 0.47 [-0.19 to 1.13]
  IADL Baseline to 3 month with covariates | 0.70 [0.34 to 1.05] | 0.47 [0.11 to 0.83] | 0.51 [-0.12 to 1.14]
Statistical Analysis 1: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of the Basic Activities of Daily Living (BADL) subscale based on contrasts between two groups at baseline to six months from mixed model ANOVA with an unstructured covariance structure; Test type: Superiority; p = 0.326, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 0.99; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.25 to 0.74] — Difference between the BADL changes (EX+T - EX+P)
Statistical Analysis 2: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.587, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -0.54; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.87 to 0.49] — Difference between the BADL changes (EX+T - EUC)
Statistical Analysis 3: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.213, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -1.25; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-1.12 to 0.25] — Difference between the BADL changes (EX+P - EUC)
Statistical Analysis 4: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of the Basic Activities of Daily Living (BADL) subscale based on contrasts between two groups at baseline to six months from mixed model ANOVA with a Toeplitz covariance structure in the model with covariates; Test type: Superiority; p = 0.410, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.83; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.32 to 0.78] — Difference between the BADL changes (EX+T - EX+P)
Statistical Analysis 5: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 4]; Test type: Superiority; p = 0.527, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -0.63; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.99 to 0.51] — Difference between the BADL changes (EX+T - EUC)
Statistical Analysis 6: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 4]; Test type: Superiority; p = 0.219, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -1.23; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.23 to 0.28] — Difference between the BADL changes (EX+P - EUC)
Statistical Analysis 7: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of the Basic Activities of Daily Living (BADL) subscale based on contrasts between two groups at baseline to three months from mixed model ANOVA with an unstructured covariance structure; Test type: Superiority; p = 0.355, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 0.93; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.25 to 0.69] — Difference between the BADL changes (EX+T - EX+P)
Statistical Analysis 8: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 7]; Test type: Superiority; p = 0.554, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -0.59; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.88 to 0.47] — Difference between the BADL changes (EX+T - EUC)
Statistical Analysis 9: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 7]; Test type: Superiority; p = 0.219, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -1.24; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.10 to 0.26] — Difference between the BADL changes (EX+P - EUC)
Statistical Analysis 10: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of the Basic Activities of Daily Living (BADL) subscale based on contrasts between two groups at baseline to three months from mixed model ANOVA with a Toeplitz covariance structure in the model with covariates; Test type: Superiority; p = 0.345, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.95; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.24 to 0.68] — Difference between the BADL changes (EX+T - EX+P)
Statistical Analysis 11: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 10]; Test type: Superiority; p = 0.494, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -0.69; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.88 to 0.43] — Difference between the BADL changes (EX+T - EUC)
Statistical Analysis 12: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 10]; Test type: Superiority; p = 0.180, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -1.35; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-1.11 to 0.21] — Difference between the BADL changes (EX+P - EUC)
Statistical Analysis 13: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of the Instrumental Activities of Daily Living (IADL) subscale based on contrasts between two groups at baseline to six months from mixed model ANOVA with an unstructured covariance structure; Test type: Superiority; p = 0.693, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -0.4; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.75 to 0.50] — Difference between the changes of IADL of EX+T - EX+P
Statistical Analysis 14: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 13]; Test type: Superiority; p = 0.327, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -0.98; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.27 to 0.43] — Difference between the IADL changes (EX+T - EUC)
Statistical Analysis 15: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 13]; Test type: Superiority; p = 0.493, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = -0.69; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-1.15 to 0.56] — Difference between the IADL changes (EX+P - EUC)
Statistical Analysis 16: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of the Instrumental Activities of Daily Living (IADL) subscale based on contrasts between two groups at baseline to six months from mixed model ANOVA with an Autoregressive (1) covariance structure in the model with covariates; Test type: Superiority; p = 0.698, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -0.39; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.72 to 0.49] — Difference between the IADL changes (EX+T - EX+P)
Statistical Analysis 17: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 16]; Test type: Superiority; p = 0.404, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -0.84; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-1.17 to 0.47] — Difference between the IADL changes (EX+T - EUC)
Statistical Analysis 18: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 16]; Test type: Superiority; p = 0.585, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -0.55; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-1.06 to 0.60] — Difference between the IADL changes (EX+P - EUC)
Statistical Analysis 19: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of the Instrumental Activities of Daily Living (IADL) subscale based on contrasts between two groups at baseline to three months from mixed model ANOVA with an unstructured covariance structure; Test type: Superiority; p = 0.399, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 0.85; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.31 to 0.76] — Difference between IADL changes (EX+T - EX+P)
Statistical Analysis 20: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 19]; Test type: Superiority; p = 0.554, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 0.59; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.53 to 0.98] — Difference between the IADL changes (EX+T - EUC)
Statistical Analysis 21: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 19]; Test type: Superiority; p = 0.998, Mixed Models Analysis — Unadjusted p-value; t (df, 112) = 0; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.76 to 0.76] — Difference between the IADL changes (EX+P - EUC)
Statistical Analysis 22: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of the Instrumental Activities of Daily Living (IADL) subscale based on contrasts between two groups at baseline to three months from mixed model ANOVA with an Autoregressive (1) covariance structure in the model with covariates; Test type: Superiority; p = 0.378, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.88; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.28 to 0.73] — Difference between the IADL changes (EX+T - EX+P)
Statistical Analysis 23: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 22]; Test type: Superiority; p = 0.608, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.51; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.53 to 0.91] — Difference between the IADL changes (EX+T - EUC)
Statistical Analysis 24: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 7, analysis 22]; Test type: Superiority; p = 0.915, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -0.11; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.76 to 0.69] — Difference between the IADL changes (EX+P - EUC)

8. Secondary Outcome: Change in Functional Status Questionnaire (FSQ) Total Score
Description: The Functional Status Questionnaire (FSQ) is a self-reported measure asking about the amount of difficulty a participant experienced when performing daily tasks in the previous 4 weeks. There are a total of 6 subscales, but only the basic ADL and Intermediate ADL were used in the STEP-HI study for a total of 9 items. Scores range from 0 (high amount of difficulty completing tasks) to 36 (no difficulty completing tasks). Per the protocol: In addition to the primary analysis (unadjusted baseline to 6 month comparison), statistical contracts were evaluated to determine if there was significant between-group differences in the change from baseline to 3 months and additional analysis of covariance were performed to adjust for baseline values and covariates that differed across groups at baseline.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 53 | 51 | 18
units on a scale
  Unadjusted baseline to 6 month | 2.04 [0.75 to 3.33] | 1.55 [0.24 to 2.49] | 3.00 [0.84 to 5.16]
  Baseline to 6 month with covariates | 2.02 [0.67 to 3.38] | 1.56 [0.18 to 2.94] | 3.06 [0.81 to 5.31]
  Unadjusted baseline to 3 month | 1.83 [0.72 to 2.94] | 1.35 [0.22 to 2.49] | 1.95 [-0.02 to 3.92]
  Baseline to 3 month with covariates | 1.83 [0.73 to 2.93] | 1.35 [0.24 to 2.47] | 1.99 [0.06 to 3.92]
Statistical Analysis 1: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to six months from mixed model ANOVA with a Toeplitz covariance structure; Test type: Superiority; p = 0.602, Mixed Models Analysis — Unadjusted p-value; t (df, 234) = 0.52; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-1.36 to 2.33] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 2: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.454, Mixed Models Analysis — Unadjusted p-value; t (df, 234) = -0.75; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-3.48 to 1.56] — Difference between the changes (EX+T - EUC)
Statistical Analysis 3: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.262, Mixed Models Analysis — Unadjusted p-value; t (df, 234) = -1.13; Mean Difference (Final Values) = -1.45, 95% CI 2-sided [-3.98 to 1.09] — Difference between the changes (EX+P - EUC)
Statistical Analysis 4: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.639, Mixed Models Analysis — Unadjusted p-value; t (df, 234) = 0.47; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-1.47 to 2.40] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 5: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.438, Mixed Models Analysis — Unadjusted p-value; t (df, 234) = -0.78; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-3.66 to 1.59] — Difference between the changes (EX+T - EUC)
Statistical Analysis 6: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.265, Mixed Models Analysis — Unadjusted p-value; t (df, 234) = -1.12; Mean Difference (Final Values) = -1.50, 95% CI 2-sided [-4.14 to 1.14] — Difference between the changes (EX+P - EUC)
Statistical Analysis 7: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to three months from mixed model ANOVA with a Toeplitz covariance structure; Test type: Superiority; p = 0.555, Mixed Models Analysis — Unadjusted p-value; t (df, 234) = 0.59; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [-1.11 to 2.07] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 8: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 8, analysis 7]; Test type: Superiority; p = 0.917, Mixed Models Analysis — Unadjusted p-value; t (df, 234) = -0.10; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-2.39 to 2.15] — Difference between the changes (EX+T - EUC)
Statistical Analysis 9: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 8, analysis 7]; Test type: Superiority; p = 0.606, Mixed Models Analysis — Unadjusted p-value; t (df, 234) = -0.52; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-2.87 to 1.68] — Difference between the changes (EX+P - EUC)
Statistical Analysis 10: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 1, analysis 10]; Test type: Superiority; p = 0.549, Mixed Models Analysis — Unadjusted p-value; t (df, 234) = 0.60; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [-1.09 to 2.04] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 11: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 10]; Test type: Superiority; p = 0.887, Mixed Models Analysis — Unadjusted p-value; t (df, 234) = -0.14; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-2.38 to 2.06] — Difference between the changes (EX+T - EUC)
Statistical Analysis 12: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 1, analysis 10]; Test type: Superiority; p = 0.574, Mixed Models Analysis — Unadjusted p-value; t (df, 234) = -0.56; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-2.87 to 1.59] — Difference between the changes (EX+P - EUC)

9. Secondary Outcome: Change in Hip Rating Questionnaire Total Score
Description: The Hip Rating Questionnaire (HRQ) Standardized is a 14-item scale with weighted questions regarding quality of life (pain level and ability to walk) and function (ability to use stairs, put on socks/shoes, use public transportation, bathe, shop, do housework, and get in and out of a chair/bed) related to the hip fracture event. The scale scores range from 16 to 100. Higher scores are associated with less pain, higher function, and better quality of life. Per the protocol: In addition to the primary analysis (unadjusted baseline to 6 month comparison), statistical contracts were evaluated to determine if there was significant between-group differences in the change from baseline to 3 months and additional analysis of covariance were performed to adjust for baseline values and covariates that differed across groups at baseline.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 53 | 51 | 18
units on a scale
  Unadjusted baseline to 6 month | 8.51 [5.62 to 11.41] | 7.55 [4.58 to 10.53] | 6.01 [1.07 to 10.94]
  Baseline to 6 month with covariates | 8.48 [5.59 to 11.37] | 7.61 [4.64 to 10.57] | 6.01 [1.08 to 10.94]
  Unadjusted baseline to 3 month | 6.52 [3.65 to 9.40] | 5.98 [3.04 to 8.91] | 4.25 [-0.89 to 9.40]
  Baseline to 3 month with covariates | 6.52 [3.65 to 9.39] | 5.98 [3.05 to 8.90] | 4.63 [-0.48 to 9.74]
Statistical Analysis 1: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to six months from mixed model ANOVA with a Compound Symmetry covariance structure; Test type: Superiority; p = 0.649, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.46; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [-3.19 to 5.11] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 2: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.389, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.86; Mean Difference (Final Values) = 2.50, 95% CI 2-sided [-3.22 to 8.23] — Difference between the changes (EX+T - EUC)
Statistical Analysis 3: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.598, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.53; Mean Difference (Final Values) = 1.55, 95% CI 2-sided [-4.22 to 7.31] — Difference between the changes (EX+P - EUC)
Statistical Analysis 4: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to six months from mixed model ANOVA with a Compound Symmetry covariance structure in the model with covariates; Test type: Superiority; p = 0.676, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.42; Mean Difference (Final Values) = 0.88, 95% CI 2-sided [-3.26 to 5.02] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 5: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p = 0.394, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.85; Mean Difference (Final Values) = 2.48, 95% CI 2-sided [-3.24 to 8.19] — Difference between the changes (EX+T - EUC)
Statistical Analysis 6: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p = 0.585, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.55; Mean Difference (Final Values) = 1.60, 95% CI 2-sided [-4.15 to 7.35] — Difference between the changes (EX+P - EUC)
Statistical Analysis 7: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to three months from mixed model ANOVA with a Compound Symmetry covariance structure; Test type: Superiority; p = 0.794, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.26; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-3.56 to 4.65] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 8: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 9, analysis 7]; Test type: Superiority; p = 0.449, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.76; Mean Difference (Final Values) = 2.27, 95% CI 2-sided [-3.62 to 8.16] — Difference between the changes (EX+T - EUC)
Statistical Analysis 9: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 9, analysis 7]; Test type: Superiority; p = 0.567, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.57; Mean Difference (Final Values) = 1.72, 95% CI 2-sided [-4.20 to 7.64] — Difference between the changes (EX+P - EUC)
Statistical Analysis 10: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to three months from mixed model ANOVA with a Compound Symmetry covariance structure in the model with covariates; Test type: Superiority; p = 0.794, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.26; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-3.56 to 4.65] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 11: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 9, analysis 10]; Test type: Superiority; p = 0.526, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.64; Mean Difference (Final Values) = 1.89, 95% CI 2-sided [-3.97 to 7.75] — Difference between the changes (EX+T - EUC)
Statistical Analysis 12: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 9, analysis 10]; Test type: Superiority; p = 0.654, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.45; Mean Difference (Final Values) = 1.34, 95% CI 2-sided [-4.55 to 7.23] — Difference between the changes (EX+P - EUC)

10. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health
Description: Patient-Reported Outcomes Measurement Information System (PROMIS®) Global Health instrument is a 10 item self report questionnaire used to measure overall quality of life using 2 summary scores: Physical and Mental Health. Each summary score is standardized to the general population, with the average T-score for the US population being 50 and standard deviation of 10. Each individual participant T-score from Baseline was subtracted from Month 6 T-score to represent change over the length of the study. Higher scores represent larger increases in Physical and Mental Health. Per the protocol: In addition to the primary analysis (unadjusted baseline to 6 month comparison), statistical contracts were evaluated to determine if there was significant between-group differences in the change from baseline to 3 months and additional analysis of covariance were performed to adjust for baseline values and covariates that differed across groups at baseline.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 53 | 51 | 18
T-score
  Physical Health - Unadjusted baseline to 6 month | 1.89 [0.25 to 3.52] | 1.25 [-0.43 to 2.94] | 4.07 [1.29 to 6.85]
  Physical Health - Baseline to 6 month with covariates | 1.88 [0.03 to 3.72] | 1.24 [-0.65 to 3.13] | 4.03 [0.92 to 7.13]
  Physical Health - Unadjusted baseline to 3 month | 2.61 [1.01 to 4.22] | 1.09 [-0.54 to 2.73] | 1.17 [-1.72 to 4.06]
  Physical Health - Baseline to 3 month with covariates | 2.61 [1.00 to 4.23] | 1.09 [-0.55 to 2.74] | 1.26 [-1.60 to 4.12]
  Mental Health - Unadjusted baseline to 6 month | 1.55 [-0.25 to 3.34] | -0.76 [-2.61 to 1.08] | 1.58 [-1.39 to 4.56]
  Mental Health - Baseline to 6 month with covariates | 1.47 [-0.22 to 3.16] | -0.69 [-2.42 to 1.04] | 1.93 [-0.90 to 4.77]
  Mental Health - Unadjusted baseline to 3 month | 1.59 [0.09 to 3.08] | 0.01 [-1.53 to 1.55] | 2.19 [-0.46 to 4.84]
  Mental Health - Baseline to 3 month with covariates | 1.59 [0.12 to 3.05] | 0.00 [-1.51 to 1.50] | 2.28 [-0.32 to 4.88]
Statistical Analysis 1: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of Physical Health Domain based on contrasts between two groups at baseline to six months from mixed model ANOVA with a Heterogeneous Toeplitz covariance structure; Test type: Superiority; p = 0.597, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.53; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-1.72 to 2.98] — Difference between the changes (EX+T - EX+P) on Physical Health domain
Statistical Analysis 2: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.184, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -1.33; Mean Difference (Final Values) = -2.18, 95% CI 2-sided [-5.41 to 1.04] — Difference between the changes (EX+T - EUC) on Physical Health domain
Statistical Analysis 3: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.089, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -1.71; Mean Difference (Final Values) = -2.82, 95% CI 2-sided [-6.07 to 0.44] — Difference between the changes (EX+P - EUC) on Physical Health domain
Statistical Analysis 4: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of Physical Health Domain based on contrasts between two groups at baseline to six months from mixed model ANOVA with a Heterogeneous Toeplitz covariance structure in the model with covariates; Test type: Superiority; p = 0.635, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.47; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [-2.01 to 3.28] — Difference in the changes (EX+T - EX+P)
Statistical Analysis 5: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 4]; Test type: Superiority; p = 0.242, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -1.17; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-5.76 to 1.46] — Difference between the changes (EX+T - EUC)
Statistical Analysis 6: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 4]; Test type: Superiority; p = 0.132, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -1.51; Mean Difference (Final Values) = -2.79, 95% CI 2-sided [-6.42 to 0.85] — Difference between the changes (EX+P - EUC)
Statistical Analysis 7: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of Physical Health Domain based on contrasts between two groups at baseline to three months from mixed model ANOVA with a Heterogeneous Toeplitz covariance structure; Test type: Superiority; p = 0.193, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 1.31; Mean Difference (Final Values) = 1.52, 95% CI 2-sided [-0.77 to 3.81] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 8: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.390, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.86; Mean Difference (Final Values) = 1.44, 95% CI 2-sided [-1.86 to 4.75] — Difference between the changes (EX+T - EUC)
Statistical Analysis 9: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.965, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -0.04; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-3.39 to 3.25] — Difference between the changes (EX+P - EUC)
Statistical Analysis 10: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of Physical Health Domain based on contrasts between two groups at baseline to three months from mixed model ANOVA with a Heterogeneous Toeplitz covariance structure in the model with covariates; Test type: Superiority; p = 0.195, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 1.30; Mean Difference (Final Values) = 1.52, 95% CI 2-sided [-0.79 to 3.82] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 11: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 10]; Test type: Superiority; p = 0.418, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = 0.81; Mean Difference (Final Values) = 1.35, 95% CI 2-sided [-1.93 to 4.63] — Difference between the changes (EX+T - EUC)
Statistical Analysis 12: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 10]; Test type: Superiority; p = 0.921, Mixed Models Analysis — Unadjusted p-value; t (df, 233) = -0.10; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-3.46 to 3.13] — Difference between the changes (EX+P - EUC)
Statistical Analysis 13: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of Mental Health Domain based on contrasts between two groups at baseline to six months from mixed model ANOVA with a Heterogeneous AR Autoregressive (1) covariance structure; Test type: Superiority; p = 0.078, Mixed Models Analysis — Unadjusted p-value; t (df, 232) = 1.77; Mean Difference (Final Values) = 2.31, 95% CI 2-sided [-0.26 to 4.88] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 14: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 13]; Test type: Superiority; p = 0.982, Mixed Models Analysis — Unadjusted p-value; t (df, 232) = -0.02; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-3.51 to 3.43] — Difference between the changes (EX+T - EUC)
Statistical Analysis 15: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 13]; Test type: Superiority; p = 0.187, Mixed Models Analysis — Unadjusted p-value; t (df, 232) = -1.32; Mean Difference (Final Values) = -2.35, 95% CI 2-sided [-5.85 to 1.15] — Difference between the changes (EX+P - EUC)
Statistical Analysis 16: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of Mental Health Domain based on contrasts between two groups at baseline to six months from mixed model ANOVA with a Heterogeneous AR Autoregressive (1) covariance structure in the model with covariates; Test type: Superiority; p = 0.080, Mixed Models Analysis — Unadjusted p-value; t (df, 232) = 1.76; Mean Difference (Final Values) = 2.16, 95% CI 2-sided [-0.26 to 4.58] — Difference of the changes (EX+T - EX+P)
Statistical Analysis 17: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 16]; Test type: Superiority; p = 0.781, Mixed Models Analysis — Unadjusted p-value; t (df, 232) = -0.28; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-3.76 to 2.83] — Difference between the changes (EX+T - EUC)
Statistical Analysis 18: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 16]; Test type: Superiority; p = 0.121, Mixed Models Analysis — Unadjusted p-value; t (df, 232) = -1.56; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-5.94 to 0.69] — Difference between the changes (EX+P - EUC)
Statistical Analysis 19: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of Mental Health Domain based on contrasts between two groups at baseline to three months from mixed model ANOVA with a Heterogeneous AR Autoregressive (1) covariance structure; Test type: Superiority; p = 0.148, Mixed Models Analysis — Unadjusted p-value; t (df, 232) = 1.45; Mean Difference (Final Values) = 1.58, 95% CI 2-sided [-0.57 to 3.73] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 20: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 19]; Test type: Superiority; p = 0.699, Mixed Models Analysis — Unadjusted p-value; t (df, 232) = -0.39; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-3.64 to 2.45] — Differences between the changes (EX+T - EUC)
Statistical Analysis 21: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 19]; Test type: Superiority; p = 0.163, Mixed Models Analysis — Unadjusted p-value; t (df, 232) = -1.4; Mean Difference (Final Values) = -2.18, 95% CI 2-sided [-5.24 to 0.89] — Difference in the changes (EX+P - EUC)
Statistical Analysis 22: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison of Mental Health Domain based on contrasts between two groups at baseline to three months from mixed model ANOVA with a Heterogeneous AR Autoregressive (1) covariance structure in the model with covariates; Test type: Superiority; p = 0.137, Mixed Models Analysis — Unadjusted p-value; t (df, 232) = 1.49; Mean Difference (Final Values) = 1.59, 95% CI 2-sided [-0.51 to 3.69] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 23: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 22]; Test type: Superiority; p = 0.648, Mixed Models Analysis — Unadjusted p-value; t (df, 232) = -0.46; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-3.68 to 2.29] — Difference between the changes (EX+T - EUC)
Statistical Analysis 24: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 10, analysis 22]; Test type: Superiority; p = 0.135, Mixed Models Analysis — Unadjusted p-value; t (df, 232) = -1.50; Mean Difference (Final Values) = -2.28, 95% CI 2-sided [-5.29 to 0.72] — Difference between the changes (EX+P - EUC)

11. Secondary Outcome: Change in Bone Mineral Density (BMD) of the Non-fractured Proximal Femur
Description: Bone mineral density (BMD) measured by dual x-ray absorptiometry (DXA) of the non-fractured proximal femur in participants without hardware in the contralateral hip. Baseline DXA scans were completed prior to the first administration of study drug. All scans were completed prior to exercise or 1-RM measurements if scheduled for the same day. DXA scans were reviewed for quality control, proper positioning, and artifacts centrally. Per the protocol: In addition to the primary analysis (unadjusted baseline to 6 month comparison), additional analysis of covariance were performed to adjust for baseline values and covariates that differed across groups at baseline. DXA was not performed at 3 months.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: g/cm^2
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 53 | 51 | 18
g/cm^2
  Unadjusted baseline to 6 month | -0.008 [-0.054 to 0.038] | -0.001 [-0.047 to 0.046] | -0.021 [-0.104 to 0.062]
  Baseline to 6 month with covariates | -0.002 [-0.009 to 0.006] | 0.001 [-0.007 to 0.008] | 0.000 [-0.013 to 0.014]
Statistical Analysis 1: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); Comparison based on contrasts between two groups at baseline to six months from mixed model ANOVA with an Autoregressive AR(1) covariance structure; Test type: Superiority; p = 0.821, Mixed Models Analysis — Unadjusted p-value; t (df, 92) = -0.23; Mean Difference (Final Values) = -0.008, 95% CI 2-sided [-0.073 to 0.058] — Difference between the changes (EX+T - EX+P)
Statistical Analysis 2: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.789, Mixed Models Analysis — Unadjusted p-value; t (df, 92) = 0.27; Mean Difference (Final Values) = 0.013, 95% CI 2-sided [-0.082 to 0.108] — Difference between the changes (EX+T - EUC)
Statistical Analysis 3: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.672, Mixed Models Analysis — Unadjusted p-value; t (df, 92) = 0.42; Mean Difference (Final Values) = 0.020, 95% CI 2-sided [-0.075 to 0.116] — Difference between the changes (EX+P - EUC)
Statistical Analysis 4: Comparison: Exercise + Testosterone (EX + T) vs Exercise + Placebo (EX + P); [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p = 0.703, Mixed Models Analysis — Unadjusted p-value; t (df, 92) = -0.38; Mean Difference (Final Values) = -0.002, 95% CI 2-sided [-0.013 to 0.009]; Difference between the changes (EX+T - EX+P)
Statistical Analysis 5: Comparison: Exercise + Testosterone (EX + T) vs Enhanced Usual Care (EUC); [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p = 0.803, Mixed Models Analysis — Unadjusted p-value; t (df, 92) = -0.25; Mean Difference (Final Values) = -0.002, 95% CI 2-sided [-0.017 to 0.014]; Difference between the changes (EX+T - EUC)
Statistical Analysis 6: Comparison: Exercise + Placebo (EX + P) vs Enhanced Usual Care (EUC); [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p = 0.991, Mixed Models Analysis — Unadjusted p-value; t (df, 92) = 0.01; Mean Difference (Final Values) = 0.000, 95% CI 2-sided [-0.015 to 0.016]; Difference between the changes (EX+P - EUC)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization until 30 days after the participant's final assessment visit (either 6 months after randomization or early withdrawal) or any subsequent event believed to be reasonably related to participation in the study. After consent, but prior to randomization, adverse events that were a direct result of study procedures or occurred while the participant was under study staff supervision were also collected.
Description: At each monthly visit, participants were asked specific questions to elicit adverse events. Participants were asked to keep a daily log of falls, illnesses, and doctor's appointments to assist with adverse events assessment and recollection. Safety labs were drawn at baseline, Month 3, and Month 6. Any spontaneous report or visualized incident was also reported.
Arm/Group | Exercise + Testosterone (EX + T) | Exercise + Placebo (EX + P) | Enhanced Usual Care (EUC)
All-Cause Mortality (participants affected / at risk) | 1/55 | 0/54 | 0/20
Serious Adverse Events (participants affected / at risk) | 7/54 | 3/55 | 1/20
Other Adverse Events (participants affected / at risk) | 36/54 | 24/55 | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise + Testosterone (EX + T) (N=54) | Exercise + Placebo (EX + P) (N=55) | Enhanced Usual Care (EUC) (N=20)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ruptured diverticulum of colon (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Large intestine perforation
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Kidney fibrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Renal scarring
Medical device complication (General disorders) | 0 (0) | 1 (1) | 0 (0) — Loosening of stabilization hardware of hip fracture repair
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Buttock pain
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Sigmoid diverticulosis
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting bile (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise + Testosterone (EX + T) (N=54) | Exercise + Placebo (EX + P) (N=55) | Enhanced Usual Care (EUC) (N=20)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (7) | 1 (2) | 0 (0)
Edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema peripheral (General disorders) | 0 (0) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (5) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 7 (7) | 2 (3) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Blood Calcium increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 3 (5) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 3 (3) | 2 (2) — 2 additional participants complained of arthralgia after screening, but did not randomize.
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 2 (2) — One additional participant complained of back pain after screening, but did not randomize.
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Bunion
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (8) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 3 (8) | 0 (0)
Hypotension (Vascular disorders) | 4 (6) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT02938923/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT02938923/ICF_002.pdf